CLINICAL TRIAL: NCT02105805
Title: Intentional Weight Loss as Treatment in Obese Patients With Ischaemic Heart Disease
Brief Title: Weight Loss as Treatment in Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-01-clinnutr
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Heart Failure
Keywords: intention weight loss; heart failure; 6-minute walk test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low energy diet (Experimental): low energy diet treatment
  Interventions: Behavioral: Dietetic group sessions
- Nordic recommendation (Active Comparator): Nordic recommendation, no restrictions on energy
  Interventions: Behavioral: Dietetic group sessions

INTERVENTIONS:
Behavioral: Dietetic group sessions — Group sessions to improve dietary adherence

SUMMARY:
30 obese moderate-to-severe heart failure patients will be randomized to intervention or control in groups of 5-10 subjects.

All will receive dietetic advice according to randomization and according to the European Heart Association.

Intervention subjects will initiate with 8 weeks low energy diet, 800-1000 kcal/d by formula diet and subsequent four weeks reintroduction to regular foods supplying 1200 kcal/d substituting two daily meals with formula meal replacement.

Control subjects are advised to follow the Nordic Nutrition Recommendations.

Patients will be monitored by blood sampling and assessed by change in physical performance.

ELIGIBILITY:
Inclusion Criteria:

* bmi >30
* heart failure, moderate to severe, new york heart association II og III
* stable disease
* age >18 years
* out-patients
* perform a six minutes walk test
* given consent

Exclusion Criteria:

* unstable disease
* insulin treated diabetes
* pregnancy or lactating
* unstable weight past 6 months (+- 10 kg)
* planned procedures in the time of intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in six minute walk test from baseline to week 16 (end of study) | weeks 0 and 16
  Performance measure

SECONDARY OUTCOMES:
Change in lipid status from baseline to week 16 (end of study). | weeks 0,1,2,4,6,8,10,12,14,16
  Blood sample and analyses for lipids